CLINICAL TRIAL: NCT06307171
Title: Human Leishmaniasis: Antigen Recognition Pattern and Study of New Potential Biomarkers
Acronym: LeishmARPs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-11
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Leishmaniasis
MeSH Terms: conditions — Leishmaniasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Leishmaniasis cases (Other): Archived, cryo-preserved or prospectively collected samples from patients with clinically or laboratory confirmed leishmaniasis
  Interventions: Diagnostic Test: In-house Western blot, specific for Leishmania
- Community Controls (Other): Sera from uninfected subject archived, cryo-preserved serum sample,stored at the Tropica Biobank at the DITM, IRCCS Sacro Cuore Don Calabria Hospital, Negrar (Vr), from subjects from Italy and from Africa with negative results to two serological test for leishmaniasis. Archived, cryo-preserved serum sample from subjects with a confirmed diagnosis of Chagas' diseases, TB, leprosy, and malaria stored at the Tropica Biobank at the DITM, IRCCS Sacro Cuore Don Calabria Hospital, Negrar, Verona.
  Interventions: Diagnostic Test: In-house Western blot, specific for Leishmania
- Validation CONTROLS (VC) (Other): Serum samples stored in Tropica Biobank at the DITM from subjects that have been clinically diagnosed with Chagas's disease (n=15), or TB (n=15), or malaria (n=15) or leprosy (n=5).
  Interventions: Diagnostic Test: In-house Western blot, specific for Leishmania

INTERVENTIONS:
Diagnostic Test: In-house Western blot, specific for Leishmania — Sample will be collected at the collaborating centres and at the DITM, if not already stored at -80°C. The samples will be delivered to the DITM. For the CONTROL groups, two serological tests for Leishmaniasis, based on different antigenic fraction, will be performed on serum samples.
  Different strains of Leishmania infantum and Leishmania donovani will be cultivated axenically at the DITM.
  Whole soluble fraction of promastigote (WSF), the whole membrane protein fraction (WMF) and the whole soluble fraction secreted by promastigotes (WSFe) of Leishmania spp. will be obtained and the ARPs from WSF, WMF and WSFe, of each Leishmania will be checked trough Western-blot analysis testing at a final dilution of 1/100 each serum sample. The predominant bands detected by Western-blot analysis will be identified by SDS-PAGE separation. Selected bands, corresponding to the immunogenic bands, will be excised, digested and identified with Mass Spectrometry analysis.

SUMMARY:
This is an exploratory experimental multicentre study on archived serum samples and on prospectively collected serum samples and blood samples.

General objectives of the study are: to identify specific biomarkers in order to develop more accurate serological tests for the screening of Leishmania infections that does not present cross-reaction with other infectious diseases; to unveil the Antigen Recognition Patterns (ARPs) of Leishmania infection in humans; to verify whether the ARPs and the new biomarkers are common to different Leishmania infantum strains isolated in Italy as well as in other part of the World and to different strains of L. donovani isolated in Sudan as well as in other part of the World and discard any possible cross reaction with other infectious diseases such as Chagas, TB, leprosy or malaria.

ELIGIBILITY:
CASES:

Inclusion criteria:

* Leishmania positive patient from Italy (n=30) and from Sudan (n=30);
* patient with a clinically or laboratory confirmed diagnosis of leishmaniasis;
* signed informed consent (criteria not applied in case of samples stored at the Tropica Biobank at the DITM)
* being clinically classified as leishmaniasis patient by an experienced clinician or being laboratory confirmed as leishmaniasis patients, giving positive to at least two different serological tests or to a molecular test for Leishmania sp.
* adult subjects (equal or older than 18 years)

Exclusion criteria:

* lack of the necessary data and/or of biological samples
* subjects younger than 18 years

COMMUNITY CONTROLS:

Inclusion criteria:

* Cryo-preserved serum samples stored at the Tropica Biobank at the DITM , IRCCS Sacro Cuore Don Calabria Hospital, Negrar (Vr), from subject from Italy (n=30) and from Africa (n=30) with no infection due by Leishmania spp.
* signed informed consent to Tropica Biobank
* adult subjects (equal or older than 18 years)
* being negative to two different serological tests for leishmaniasis

Exclusion criteria:

* subjects younger than 18 years
* being positive to one serological tests for leishmaniasis.

VALIDATION CONTROLS (VC):

Inclusion criteria:

* serum samples stored in Tropica Biobank at the DITM from subjects that have been clinically diagnosed with Chagas's disease, or TB, or malaria or leprosy.
* informed consent signed to Tropical Biobank
* adult subjects (equal or older than 18 years)
* being negative to two different serological tests for leishmaniasis.
* being clinically diagnosed with Chagas disease or TB, or malaria or leprosy

Exclusion criteria:

* younger than 18 years
* positive result to one serological test for leishmaniasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Biomarkers from Leishmania spp | Baseline
  Presence/Absence of a reactive immunogenic band or a pattern of reactive immunogenic bands in an in-house Western blot, specific for Leishmania cases respect to negative controls.

SECONDARY OUTCOMES:
ARPs in different Leishmania infantum and L. donovani strains | Baseline
  Presence/Absence of a common or differential reactive immunogenic band/pattern in different Leishmania infantum and Leishmania donovani strains from different geographical areas.
Cross reaction | Baseline
  Presence/Absence of cross-reaction of the identified immunogenic bands, testing serum samples of patients with malaria or TB or leprosy or Chagas' disease

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Sacro Cuore Don Calabria hospital, Negrar, Verona, Italy